CLINICAL TRIAL: NCT07402135
Title: Fecal Noninvasive Biomarkers Oriented Control Versus Usual Care Strategy in Ulcerative Colitis: A Multicenter, Open-Label, Randomized, Parallel Controlled Clinical Trial
Brief Title: Fecal Noninvasive Biomarkers Oriented Control Versus Usual Care Strategy in Ulcerative Colitis
Acronym: FOCUS-UC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Qilu Hospital of Shandong University (Qingdao) (Other); Dezhou Hospital Qilu Hospital of Shandong University (Other); Weihai Municipal Hospital (Other); Jining First People's Hospital (Other); Zaozhuang Municipal Hospital (Other); Liaocheng People's Hospital (Other); Weifang People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QILUGI-002
Record Dates: First submitted 2025-07-30; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Noninvasive Biomarkers; Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tight Control (TC) Strategy (Experimental): Fecal calprotectin (FC) and FIT measured at Weeks 0, 12, 24, 36.
  Action: Preemptive therapy escalation based on preset thresholds (FC >250 μg/g or FIT >100 ng/mL) using the FOCUS-UC Ladder:
  Level 0: Current maintenance therapy. Level 1: Optimize current therapy (e.g., dose increase, TDM-guided adjustment). Level 2: Add combination therapy (e.g., biologics + immunomodulators). Level 3: Switch to advanced therapy (different mechanism). Level 4: Study withdrawal (treatment failure).
  Interventions: Procedure: Preemptive therapy escalation based on preset thresholds (FC >250 μg/g or FIT >100 ng/mL) using the FOCUS-UC Ladder:
- Conventional Management (CM) Strategy (Placebo Comparator)
  Interventions: Procedure: Therapy adjustment only upon clinical relapse (pMS increase ≥2 + rectal bleeding score ≥1).

INTERVENTIONS:
Procedure: Preemptive therapy escalation based on preset thresholds (FC >250 μg/g or FIT >100 ng/mL) using the FOCUS-UC Ladder: — Preemptive therapy escalation based on preset thresholds (FC >250 μg/g or FIT >100 ng/mL) using the FOCUS-UC Ladder:
  Level 0: Current maintenance therapy. Level 1: Optimize current therapy (e.g., dose increase, TDM-guided adjustment). Level 2: Add combination therapy (e.g., biologics + immunomodulators). Level 3: Switch to advanced therapy (different mechanism). Level 4: Study withdrawal (treatment failure).
  Arms: Tight Control (TC) Strategy
Procedure: Therapy adjustment only upon clinical relapse (pMS increase ≥2 + rectal bleeding score ≥1). — Therapy adjustment only upon clinical relapse (pMS increase ≥2 + rectal bleeding score ≥1).
  Arms: Conventional Management (CM) Strategy

SUMMARY:
Design: Multicenter, Open-Label, Randomized, Parallel Controlled Allocation: 1:1 Randomization Masking: Open-label (outcome assessors blinded for endoscopy) Primary Purpose: Treatment Strategy Evaluation Phase: Phase IV (Post-Marketing Surveillance)

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed UC diagnosis ≥6 months.
2. Clinical remission: Partial Mayo Score (pMS) ≤2, with stool frequency and rectal bleeding subscores ≤1.
3. Endoscopic remission (MES ≤1) confirmed by colonoscopy within 12 weeks pre-screening.
4. Stable maintenance therapy (5-ASA, immunomodulators, biologics, or JAK inhibitors) ≥8 weeks.
5. Written informed consent.

Exclusion Criteria:

1. Indeterminate colitis or Crohn's disease.
2. History of toxic megacolon, symptomatic colonic stricture, or dysplasia. Prior colectomy.
3. Systemic/local corticosteroid use within 8 weeks.
4. Active gastrointestinal infection or chronic diarrhea from non-UC causes.
5. Pregnancy, lactation, or concurrent interventional trial participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to Treatment Failure (Composite) | week 52
  Time to Treatment Failure (Composite):
  Clinical relapse (pMS increase ≥2 + rectal bleeding ≥1). Need for corticosteroids due to UC relapse. UC-related hospitalization or surgery. Endoscopic worsening (MES >1).

SECONDARY OUTCOMES:
Endoscopic remission rate (MES ≤1). | week 52

IPD SHARING:
Plan to Share IPD: No